CLINICAL TRIAL: NCT01145313
Title: Impact of Atypical Antipsychotic Therapy on Health Outcomes and Costs Among Patients With Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: CN138-582
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2010-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with Major Depressive Disorder: Patients diagnosed with MDD who are treated with antidepressants and subsequently augment with atypical antipsychotic therapy.

SUMMARY:
The primary objective is to examine changes in pre/post-augmentation healthcare costs and resource utilization in patients diagnosed with major depressive disorder (MDD) who augment their current antidepressant therapy with an atypical antipsychotic.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following criteria will be included in the study:

* aged 18 to 64 years
* diagnosis of major depressive disorder during the study timeframe (ICD 9 codes 296.2, 296.3, 311)
* evidence of at least 6 consecutive claims for traditional antidepressant therapy with a 30 day supply or at least 2 claims with a 90 day supply (consecutive defined as ≤15 days gap)
* must be continually enrolled during the study timeframe and have both medical and pharmacy benefits
* evidence of at least 4 consecutive claims for an atypical antipsychotic prescription with a 30 day supply or 2 claims with a 90 day supply (consecutive defined as ≤15 days gap)
* evidence of antidepressant therapy for at least 60 consecutive days prior to the initiation of atypical antipsychotic
* After at least a 60 day trial of traditional antidepressant medications, patient augments with an atypical antipsychotic medication for at least 4 months.

Exclusion Criteria:

Patients are excluded if they:

* have any claims for a diagnosis of schizophrenia, schizoaffective or bipolar disorder during the study period
* have Electroconvulsive therapy (ECT) during the study period
* new augmentation with mood stabilizers, L-thyroxine (T4), L-Thyronine (T3), buspirone, stimulant, or others during the post-period (table 1)
* are pregnant during the study period
* patients with Medicare or Medicaid

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population is identified as patients diagnosed with MDD who are treated with antidepressants and subsequently augment with atypical antipsychotic therapy.
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pre/post-augmentation healthcare costs and resource utilization among patients diagnosed with MDD who augment antidepressant therapy with an atypical antipsychotic. | 3 months pre- augmentation.
Pre/post-augmentation healthcare costs and resource utilization among patients diagnosed with MDD who augment antidepressant therapy with an atypical antipsychotic. | 3 months post-augmentation.

SECONDARY OUTCOMES:
A secondary post-hoc analysis may be conducted to determine differences in outcomes among patients during a longer treatment period, ie 6 month pre- and 6 month post-augmentation. | 6 month pre-augmentation
A secondary post-hoc analysis may be conducted to determine differences in outcomes among patients during a longer treatment period, ie 6 month pre- and 6 month post-augmentation. | 6 month post-augmentation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm